CLINICAL TRIAL: NCT07245264
Title: Randomized Trial Comparing Adjuvant Tranexamic Acid Versus Surgery Alone For Chronic Subdural Hematoma
Brief Title: Adjuvant Tranexamic Acid (TXA) Versus Surgery Alone for Adult Patients With Chronic Subdural Hematoma (CSDH)
Acronym: RATATA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHG-090891
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic subdural hematoma; Tranexamic acid; Neurosurgery
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard surgical treatment with adjunctive treatment with tranexamic acid (Active Comparator): Surgical evacuation with tranexamic acid. Preoperative administration of 1g IV with additional 1g administrated postoperatively. Followed by 500mg two times a day for a total of 28 days.
  Interventions: Drug: Tranexamic Acid (Cyklokapron)
- Standard surgical treatment (No Intervention): Surgically evacuation of chronic subdural hematoma without adjuntive medical therapy

INTERVENTIONS:
Drug: Tranexamic Acid (Cyklokapron) — Patients randomized to the treatment group will receive 1g of TXA pre and postoperative intravenously administrated followed by a 28 days treatment course of 500mg x2 of TXA orally
  Arms: Standard surgical treatment with adjunctive treatment with tranexamic acid

SUMMARY:
This study is an open label randomized controlled trial. Patients with a symptomatic Chronic Subdural Hematoma (CSDH) confirmed on radiological imaging, planned for surgery, age over 18, free from other intracranial pathologies and no previous intracranial surgery, will be recruited at time of admission. Patients eligible for inclusion will be randomized to receive treatment with Tranexamic acid (TXA) as an adjunct to surgery or surgery alone. Surgical evacuation will be performed using a single or double burr hole and 24 hours postoperative drainage. The primary endpoint will be recurrent hematoma requiring repeat surgery within 90 days. Secondary outcomes will be modified Rankin Scale at 90 days, EQ-5D-5L, complications and adverse events, and 90-day mortality.

DETAILED DESCRIPTION:
This study is a prospective single-center open-label randomized controlled trial (RCT) investigating whether the administration of tranexamic acid (TXA) as an adjuvant to surgery reduces the recurrence rate of chronic subdural hematoma (CSDH) compared to surgery alone.

CSDH is a frequent neurosurgical condition, especially among elderly patients, and carries a substantial risk of recurrence after surgical evacuation. Despite standardized procedures such as burr hole drainage and postoperative irrigation with 24-hour drainage, reoperation rates remain high (5-20%). There is currently a need for adjunctive therapies to reduce recurrence and improve clinical outcomes.

Tranexamic acid is a well-established antifibrinolytic agent that inhibits plasminogen activation and stabilizes blood clots. While observational studies and limited randomized trials have suggested a potential benefit of TXA in CSDH patients, conclusive evidence remains lacking.

This trial (RATATA) randomly assigns eligible adult patients with symptomatic CSDH confirmed via CT or MRI to receive either standard surgical treatment or surgery plus adjuvant TXA. Participants in the intervention arm receive a total of 2g IV TXA (1g <12h pre-op and 1g 12h post-op) and continue with oral TXA 500 mg twice daily for four weeks.

The primary endpoint is recurrence of the ipsilateral CSDH requiring repeat surgery within 90 days of the index operation. Recurrence is defined by both clinical deterioration and radiologically confirmed hematoma. Secondary endpoints include functional outcomes measured by the Modified Rankin Scale (mRS), health-related quality of life assessed using EQ-5D-5L, complication and adverse event rates, and 90-days mortality.

Imaging assessments will be conducted at baseline and during follow-up (post-operatively, week 4 and at surgeons´ discretion 12 weeks if indicated). The study also includes robust safety monitoring for thromboembolic and other TXA-related adverse events.

Randomization is stratified by age (≥60 vs. <60) and gender using a computer-generated block randomization scheme. Allocation concealment is ensured via sealed opaque envelopes, and outcomes assessors for imaging and functional scores are blinded to treatment assignment.

Sample size was calculated to detect a 12% absolute reduction in recurrence (from 18% to 6%), requiring 274 patients (137 per group) with 80% power and a two-sided alpha of 0.05, accounting for a 20% loss to follow-up.

The study follows Good Clinical Practice guidelines and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic chronic subdural hematoma confirmed on computer tomography (CT) or magnetic resonance imaging (MRI) measuring greater than 10 mm thickness.
2. Adult patient ≥18 years
3. Scheduled for single or double burr hole for evacuation.
4. No contraindication for TXA

Exclusion criteria

1. Mechanical heart valve
2. Newly diagnosed (last 12 months) pulmonary embolism, myocardial infarction, and strong indication for antithrombotic treatment
3. Intracranial surgery within last 6 months
4. Pregnancy and woman<40 years
5. Participation in any other clinical trial
6. Life expectancy of less than one year.
7. A score on the modified Rankin scale, designed to assess functional independence, of 4 or 5 (scores range from 0 [no symptoms] to 6 [death]) before the hematoma occurred.
8. Unfit for participations for any other reason as evaluated by the including physician.
9. History of severe impairment of renal function (eGFR <30ml/min or serum creatinine >150μmol/L)
10. Known hypersensitivity or allergy to TXA
11. Inability to obtain informed consent from the patient or legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of symptomatic chronic subdural hematoma requiring repeat surgery within 90 days | 90 days
  Number of patients with a radiological and clinical significant recurrent hematoma withing 90 days

SECONDARY OUTCOMES:
Functional outcome | 90 days
  Functional outcome measured with the modified Rankin Scale (mRS) score, range 0 (no symptoms) to 6 (death)
Health-related Quality Of Life | 90 days
  Change from baseline in generic health-related quality of life measured with the five dimensional EuroQol questionnaire (EQ-5D-L)
Headache | 90 days
  Change in headache intensity measured with numerical rating scale (1-10)
Complications and adverse events | 90 days
  Complications and adverse events
Mortality | 90 days
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Chandrashekhar Gendle, MD PhD, Study Chair — Postgraduate Institute of Medical Education & Research (PGIMER); Mattis A Madsbu, MD PhD, Principal Investigator — St. Olavs University Hospital, Department of Neurosurgery; Sasha Gulati, Professor, Study Chair — St. Olavs University Hospital, Department of Neurosurgery
Locations (1):
- Post Graduate Institute of Medical Education & Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No